CLINICAL TRIAL: NCT05593380
Title: The Impact of Invasive Intracranial Pressure Monitoring Guided Management on the Functional Outcomes of Patients With Supratentorial Large Volume Cerebral Hemorrhage: An Open Label, Randomized, Controlled, Multi-center Trial (BIATICH)
Brief Title: Bleeding Intracerebral Hemorrhage With Early Invasive Intracranial Pressure Monitoring Trial
Acronym: BIATICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sjnkzhangle; 2018FY100900 (Other: Ministry of Science and Technology of China)
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Hemorrhage, Hypertensive; Intracranial Hypertension; Monitoring; Critical Care; Treatment Outcome; Invasive Intracranial Pressure Monitoring; Large-volume Cerebral Hemorrhage
Keywords: Spontaneous cerebral hemorrhage; Brain Edema; Intracranial Hypertension; Massive intracerebral hemorrhage; Treatment Outcome; invasive intracranial pressure monitoring; Large-volume cerebral hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Intracranial Hypertension; Brain Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICP monitoring (Experimental): Intracranial pressure monitoring equipment enables continuous dynamic monitoring of changes in intracranial pressure values. This technology reflects sudden shifts in intracranial pressure resulting from hemorrhage and other cranial conditions, allowing for timely adjustments in the intensity of cerebral therapeutic interventions.
  Interventions: Device: Parenchymal Intracranial pressure monitor
- imaging-clinical examination (ICE) (Other): According to routine head CT imaging examinations, dynamic observations of changes in the patient's condition should be conducted. This involves closely monitoring clinical consciousness, pupil response, limb activity, and other clinical manifestations. Adjustments to the intensity of cerebral intervention should be made based on the clinical reflections of these dynamic changes.
  Interventions: Other: Treatment based on clinical and imaging observations

INTERVENTIONS:
Device: Parenchymal Intracranial pressure monitor — Treatment based on readings from Parenchymal intracranial pressure monitor.
  Other Names: Integra Life Sciences Camino Intracranial Monitor
  Arms: ICP monitoring
Other: Treatment based on clinical and imaging observations — Treatment based on clinical and imaging observations.
  Arms: imaging-clinical examination (ICE)

SUMMARY:
Spontaneous cerebral hemorrhage (SICH) is a hemorrhage caused by the rupture of a blood vessel within the brain parenchyma that is non-traumatic. Its rapid onset and dangerous condition seriously threaten human health; it accounts for about 15% of strokes and 50% of stroke-related mortality. Hunan Province is recognized as one of the high incidence areas of cerebral hemorrhage in the world; according to statistics, the direct economic loss caused by cerebral hemorrhage in Hunan Province is more than 1 billion yuan per year, which should be paid great attention. A 30-day follow-up study of large-volume cerebral hemorrhage (defined as supratentorial hemorrhage greater than 30 ml, infratentorial greater than 5 ml, and thalamus and cerebellum greater than 15 ml) found that the morbidity and mortality rate of ICH with hemorrhage of 30-60 ml was as high as 44-74%, while the morbidity and mortality rate of ICH with hemorrhage of <30 ml was 19% and that of >60 ml was 91%. According to studies, the occurrence of hematoma occupancy and malignant cerebral edema in large-volume cerebral hemorrhage can lead to secondary malignant intracranial pressure elevation and subsequent secondary brain injury, which are the main factors of high morbidity and mortality and poor prognosis in patients with large-volume cerebral hemorrhage. Clinical monitoring and management is the key to treatment, and despite aggressive surgical treatment and anti-brain edema therapy, a large number of patients progress to malignant brain edema disease, leading to poor outcomes. This study aims to conduct a multicenter clinical trial in China investigating the role of invasive intracranial pressure (ICP) monitoring in managing patients with large-volume supratentorial intracerebral hemorrhage. The trial will evaluate whether ICP-guided treatment protocols for cerebral edema improve patient outcomes and generate evidence to support the clinical application of invasive ICP monitoring in this patient population.

DETAILED DESCRIPTION:
Intracranial pressure and cerebral edema monitoring are widely employed modalities of neurological assessment in neurocritical care patients globally. However, uncertainties remain regarding the prognostic value of invasive and noninvasive intracranial pressure monitoring and cerebral edema monitoring techniques on neurological function in patients with both traumatic and non-traumatic brain injuries. Additionally, clinical practices for these modalities vary significantly in patients with extensive cerebral hemorrhage. This study aims to determine whether continuous ambulatory monitoring of intracranial pressure, administered postoperatively to patients with large-volume cerebral hemorrhage, can enhance overall prognosis by guiding adjustments in brain-specific therapeutic intensity and reducing mortality within 90 days. The study is designed as a prospective, open-label, randomized, controlled, multi-center trial with a sample size estimated based on the efficacy observed in prior research, encompassing approximately 190 cases across 15-20 clinical institutions in China experienced in treating large-volume cerebral hemorrhage. The study population consists of patients diagnosed with significant supraventricular cerebral hemorrhage (≥30 ml, based on the Coniglobus formula) via CT examination within 48 hours of symptom onset. Informed consent was obtained from patients who met the eligibility criteria. Ethical risks associated with high-volume cerebral hemorrhage were mitigated by offering surgical treatment (either open debridement flap or endoscopic hematoma removal) in accordance with established guidelines and consideration of the patients condition, the physicians judgment, and the familys preferences. Enrolled participants were randomly assigned in a 1:1 ratio to either the invasive intracranial pressure monitoring group or the imaging-clinical examination (ICE) group. All relevant research organizations and personnel will adhere to the Declaration of Helsinki and the Chinese Standards of Good Clinical Practice. This trial has received approval from the Institutional Review Board (IRB) and Ethics Committee (EC) of Xiangya Hospital, Central South University.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and Age <80 years old.
2. Diagnosed of a supratentorial spontaneous intracerebral hemorrhage.
3. Diagnosis of supratentorial large-volume cerebral hemorrhage by CT or other imaging and meeting the diagnostic criteria for large-volume cerebral hemorrhage(hemorrhage volume ≥ 30 mL of supratentorial cerebral parenchymal hematoma volume according to the Coniglobus formula on the first CT scan at onset).
4. Participants were enrolled within 48 hours of symptom onset.
5. The family signed the informed consent.

Exclusion Criteria:

1. Traumatic cerebral hemorrhage, cerebral amyloid angiopathy(CAA), secondary cerebral hemorrhage due to other specific etiologies (aneurysm, vascular malformation, smoker's disease, coagulopathy, aneurysmal stroke, vasculitis, cerebral venous thrombosis, hemorrhagic cerebral infarction, etc.)
2. The presence of fixed bilateral dilated pupils on admission, no recovery of pupils after initial dehydration treatment, and very poor survival
3. Patients with extremely unstable vital signs after admission, with extremely poor prognosis and those considered non-viable, and patients whose families have abandoned follow-up treatment
4. Patients who are pregnant or lactating.
5. Patients with bilateral temporal skin ulceration, or subcutaneous hematoma in which monitoring electrode placement cannot be implemented
6. The presence of other serious underlying diseases (intractable hypoxemia and circulatory failure with cardiopulmonary insufficiency that is difficult to correct by treatment, severe abnormal coagulation, severely reduced platelets, severe hepatic and renal insufficiency, combined neurodegenerative diseases, psychiatric diseases, autoimmune diseases, malignant tumors, thyroid diseases, etc.)
7. The patient is agitated, coughing or choking too frequently, unable to be sedated or has difficulty in handling.
8. Those with mRS score > 2 before this onset.
9. Individuals unable to complete the follow-up phase of this trial due to psychiatric, cognitive, or emotional conditions;
10. Family members decline to provide informed consent.

Exit criteria:

1. Acute onset of other life-threatening illnesses identified as the primary cause of mortality;
2. Participants who voluntarily withdraw from the study before completion;
3. Participants deemed unsuitable for the trial's monitoring protocol post-enrollment;
4. Participants requiring a modification of the treatment plan post-enrollment due to medical reasons, resulting in compromised monitoring feasibility or significant deviations in monitoring accuracy that undermine the integrity of the final analysis.

Elimination criteria：

1. Participants who failed to record any data post-enrollment;
2. Participants who did not receive per-protocol treatment post-enrollment, were discharged within 72 hours, and had their families voluntarily withdraw informed consent;
3. Participants whose invasive intracranial pressure (ICP) monitoring probes shifted and were not promptly reinserted or calibrated, leading to excessive data errors precluding analysis;
4. Participants not receiving the invasive intracranial pressure (ICP) monitoring module according to their assigned group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
mRS score on day 90 of treatment. | 90 days
  The differences between the two groups were evaluated using the modified Rankin Scale (mRS) at 90 days post-treatment. Additionally, the proportion of patients achieving functional independence, defined as an mRS score of 0-3, was calculated.

SECONDARY OUTCOMES:
Categorical shift in Modified Rankin scale | 90 days
  The modified Rankin Scale (mRS) is utilized to assess functional outcomes following intracerebral hemorrhage (ICH), with scores ranging from 0 (no symptoms) to 6 (death). The study compared mRS scores between the two groups at 14 and 90 days post-treatment, categorized as favorable (0-3) and unfavorable (4-6) outcomes. Additionally, the study investigated other mRS classifications, including good prognosis (0-2), moderate prognosis (3-4), and poor prognosis (≥5).
Neurological recovery | 14days, 90 days
  The difference value of the NIHSS between Day 14/Day 90 and the baseline.
Duration of ICU treatment | 90 days
  Time from the start of patient randomization to stable transfer out of the ICU.
GOS-E score | 90 days
  The difference value of the GOS-E between Day 90，was used to evaluate the functional outcomes after ICH.
Quality of life score (EQ-5D) | 90 days
  Generic health status evaluated by EQ-5D questionnaire at the end of the therapy.
Length of hospitalization | 90 days
  Length of stay of patients throughout the treatment period since randomization.
The incidence of serious adverse events | 90 days
  The percentage of the Severity Adverse Events within the 14 days/90 days of the therapy.
Total mortality | 90 days
  All deaths reported post-randomization will be recorded and adjudicated
Adverse Events | 90 days
  The percentage of the Adverse Events during the therapy.
Severity Adverse Event | 14 days
  The percentage of the Severity Adverse Events within the 14 days of the therapy.
Total mortality | 14 days
  All deaths reported post-randomization will be recorded and adjudicated. Deaths will be subclassified by the adjudication committee as cardiovascular or non-cardiovascular.
Adverse Events | 14 days
  The percentage of the Adverse Events during the therapy.
The incidence of adverse events That are related to treatment | 90 days
  The incidence of complications, including intracranial infections, probe displacement, recurrent intracranial hemorrhage, and skin infections, was assessed following the random grouping of patients undergoing invasive intracranial pressure (ICP) monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Le, PhD, Principal Investigator — Department of Neurology，Xiangya Hospital, Central South University
Locations (17):
- China (17):
  - The First People's Hospital of Changde City (Changde Hospital, Xiangya School of Medicine, Central South University), Changde, Hunan
  - Changsha Central Hospital, Changsha, Hunan
  - The Fourth Hospital of Changsha, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Changsha Hospital of Traditional Chinese Medicine (Changsha Eighth Hospital), Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Hunan University of Medicine General Hospital, Huaihua, Hunan
  - Xiangxi Tujia and Miao Autonomous Prefecture People's Hospital, First Affiliated Hospital of Jishou University School of Medicine, Jishou, Hunan
  - The Central Hospital of Shaoyang, Shaoyang, Hunan
  - The Central Hospital of Xiangtan, The Affiliated Hospital of Hunan University, Xiangtan, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Zhangjiajie People's Hospital, Zhangjiajie, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Chengdu Fifth Pepole's Hospital, Chengdu, Sichuan
  - Xuanwu Hospital Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116
- [Background] Bao YH, Liang YM, Gao GY, Pan YH, Luo QZ, Jiang JY. Bilateral decompressive craniectomy for patients with malignant diffuse brain swelling after severe traumatic brain injury: a 37-case study. J Neurotrauma. 2010 Feb;27(2):341-7. doi: 10.1089/neu.2009.1040. PMID 19715392
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Chesnut RM, Temkin N, Carney N, Dikmen S, Rondina C, Videtta W, Petroni G, Lujan S, Pridgeon J, Barber J, Machamer J, Chaddock K, Celix JM, Cherner M, Hendrix T; Global Neurotrauma Research Group. A trial of intracranial-pressure monitoring in traumatic brain injury. N Engl J Med. 2012 Dec 27;367(26):2471-81. doi: 10.1056/NEJMoa1207363. Epub 2012 Dec 12. PMID 23234472
- [Background] Raj R, Bendel S, Reinikainen M, Hoppu S, Laitio R, Ala-Kokko T, Curtze S, Skrifvars MB. Costs, outcome and cost-effectiveness of neurocritical care: a multi-center observational study. Crit Care. 2018 Sep 20;22(1):225. doi: 10.1186/s13054-018-2151-5. PMID 30236140
- [Background] Kumar G, Kalita J, Misra UK. Raised intracranial pressure in acute viral encephalitis. Clin Neurol Neurosurg. 2009 Jun;111(5):399-406. doi: 10.1016/j.clineuro.2009.03.004. Epub 2009 Apr 15. PMID 19372001
- [Background] Czosnyka M, Pickard JD. Monitoring and interpretation of intracranial pressure. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):813-21. doi: 10.1136/jnnp.2003.033126. PMID 15145991
- [Background] Treggiari MM, Schutz N, Yanez ND, Romand JA. Role of intracranial pressure values and patterns in predicting outcome in traumatic brain injury: a systematic review. Neurocrit Care. 2007;6(2):104-12. doi: 10.1007/s12028-007-0012-1. PMID 17522793
- [Background] Helbok R, Olson DM, Le Roux PD, Vespa P; Participants in the International Multidisciplinary Consensus Conference on Multimodality Monitoring. Intracranial pressure and cerebral perfusion pressure monitoring in non-TBI patients: special considerations. Neurocrit Care. 2014 Dec;21 Suppl 2:S85-94. doi: 10.1007/s12028-014-0040-6. PMID 25208677
- [Background] Simma B, Burger R, Falk M, Sacher P, Fanconi S. A prospective, randomized, and controlled study of fluid management in children with severe head injury: lactated Ringer's solution versus hypertonic saline. Crit Care Med. 1998 Jul;26(7):1265-70. doi: 10.1097/00003246-199807000-00032. PMID 9671379
- [Background] O'Sullivan MG, Statham PF, Jones PA, Miller JD, Dearden NM, Piper IR, Anderson SI, Housley A, Andrews PJ, Midgley S, et al. Role of intracranial pressure monitoring in severely head-injured patients without signs of intracranial hypertension on initial computerized tomography. J Neurosurg. 1994 Jan;80(1):46-50. doi: 10.3171/jns.1994.80.1.0046. PMID 8271021
- [Background] Hiler M, Czosnyka M, Hutchinson P, Balestreri M, Smielewski P, Matta B, Pickard JD. Predictive value of initial computerized tomography scan, intracranial pressure, and state of autoregulation in patients with traumatic brain injury. J Neurosurg. 2006 May;104(5):731-7. doi: 10.3171/jns.2006.104.5.731. PMID 16703877
- [Background] Ropper AH. Management of raised intracranial pressure and hyperosmolar therapy. Pract Neurol. 2014 Jun;14(3):152-8. doi: 10.1136/practneurol-2014-000811. Epub 2014 Jan 30. PMID 24481284
- [Background] Bales JW, Bonow RH, Buckley RT, Barber J, Temkin N, Chesnut RM. Primary External Ventricular Drainage Catheter Versus Intraparenchymal ICP Monitoring: Outcome Analysis. Neurocrit Care. 2019 Aug;31(1):11-21. doi: 10.1007/s12028-019-00712-9. PMID 31037639
- [Background] Aiolfi A, Khor D, Cho J, Benjamin E, Inaba K, Demetriades D. Intracranial pressure monitoring in severe blunt head trauma: does the type of monitoring device matter? J Neurosurg. 2018 Mar;128(3):828-833. doi: 10.3171/2016.11.JNS162198. Epub 2017 May 26. PMID 28548592
- [Background] Liu H, Wang W, Cheng F, Yuan Q, Yang J, Hu J, Ren G. External Ventricular Drains versus Intraparenchymal Intracranial Pressure Monitors in Traumatic Brain Injury: A Prospective Observational Study. World Neurosurg. 2015 May;83(5):794-800. doi: 10.1016/j.wneu.2014.12.040. Epub 2014 Dec 23. PMID 25541084
- [Background] Tavakoli S, Peitz G, Ares W, Hafeez S, Grandhi R. Complications of invasive intracranial pressure monitoring devices in neurocritical care. Neurosurg Focus. 2017 Nov;43(5):E6. doi: 10.3171/2017.8.FOCUS17450. PMID 29088962
- [Background] LANGFITT TW, WEINSTEIN JD, KASSELL NF, SIMEONE FA. TRANSMISSION OF INCREASED INTRACRANIAL PRESSURE. I. WITHIN THE CRANIOSPINAL AXIS. J Neurosurg. 1964 Nov;21:989-97. doi: 10.3171/jns.1964.21.11.0989. No abstract available. PMID 14238966
- [Background] Lenfeldt N, Koskinen LO, Bergenheim AT, Malm J, Eklund A. CSF pressure assessed by lumbar puncture agrees with intracranial pressure. Neurology. 2007 Jan 9;68(2):155-8. doi: 10.1212/01.wnl.0000250270.54587.71. PMID 17210899
- [Background] Andrews PJ, Citerio G. Intracranial pressure. Part one: historical overview and basic concepts. Intensive Care Med. 2004 Sep;30(9):1730-3. doi: 10.1007/s00134-004-2376-4. Epub 2004 Jul 9. No abstract available. PMID 15243684
- [Background] Miller C, Armonda R; Participants in the International Multi-disciplinary Consensus Conference on Multimodality Monitoring. Monitoring of cerebral blood flow and ischemia in the critically ill. Neurocrit Care. 2014 Dec;21 Suppl 2:S121-8. doi: 10.1007/s12028-014-0021-9. PMID 25208667
- [Background] Nag DS, Sahu S, Swain A, Kant S. Intracranial pressure monitoring: Gold standard and recent innovations. World J Clin Cases. 2019 Jul 6;7(13):1535-1553. doi: 10.12998/wjcc.v7.i13.1535. PMID 31367614
- [Background] Fernando SM, Tran A, Cheng W, Rochwerg B, Taljaard M, Kyeremanteng K, English SW, Sekhon MS, Griesdale DEG, Dowlatshahi D, McCredie VA, Wijdicks EFM, Almenawer SA, Inaba K, Rajajee V, Perry JJ. Diagnosis of elevated intracranial pressure in critically ill adults: systematic review and meta-analysis. BMJ. 2019 Jul 24;366:l4225. doi: 10.1136/bmj.l4225. PMID 31340932
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Background] Reid A, Marchbanks RJ, Burge DM, Martin AM, Bateman DE, Pickard JD, Brightwell AP. The relationship between intracranial pressure and tympanic membrane displacement. Br J Audiol. 1990 Apr;24(2):123-9. doi: 10.3109/03005369009077853. PMID 2350622
- [Background] Lou JH, Wang J, Liu LX, He LY, Yang H, Dong WW. Measurement of brain edema by noninvasive cerebral electrical impedance in patients with massive hemispheric cerebral infarction. Eur Neurol. 2012;68(6):350-7. doi: 10.1159/000342030. Epub 2012 Oct 23. PMID 23095732
- [Background] He LY, Wang J, Luo Y, Dong WW, Liu LX. Application of non-invasive cerebral electrical impedance measurement on brain edema in patients with cerebral infarction. Neurol Res. 2010 Sep;32(7):770-4. doi: 10.1179/016164109X12478302362572. Epub 2009 Sep 1. PMID 19726011
- [Background] Makarenko S, Griesdale DE, Gooderham P, Sekhon MS. Multimodal neuromonitoring for traumatic brain injury: A shift towards individualized therapy. J Clin Neurosci. 2016 Apr;26:8-13. doi: 10.1016/j.jocn.2015.05.065. Epub 2016 Jan 2. PMID 26755455
- [Background] Dallagiacoma S, Robba C, Graziano F, Rebora P, Hemphill JC, Galimberti S, Citerio G; SYNAPSE-ICU Investigators. Intracranial Pressure Monitoring in Patients With Spontaneous Intracerebral Hemorrhage: Insights From the SYNAPSE-ICU Study. Neurology. 2022 Jul 12;99(2):e98-e108. doi: 10.1212/WNL.0000000000200568. Epub 2022 May 4. PMID 35508390
- See also: Chinese Expert Consensus on Monitoring and Treatment of Spontaneous Large Volume Cerebral Hemorrhage — http://rs.yiigle.com/CN112137201709/972019.htm
- See also: An applied research on non-invasive and dynamic monitor of cerebral edema in patients after craniotomy — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDZHYX&filename=ZHCS201708016&uniplatform=NZKPT&v=OTLqMwQkzJB53apyj50gXP473ZTeWwtlkohToiHUng0eDpXbcih6qYcsaWiYBAnL
- See also: Trunk subdivision bioelectrical impedance analysis of body composition — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CMFD&dbname=CMFD2009&filename=2009064300.nh&uniplatform=NZKPT&v=AOpPQzQDMl-VJZ8H-KWRPhyaLhowckOyadDTtb6G6erEL1sKBd34MTJGx9FpqcTE
- See also: Disturbance method of electric current field and its application in impedance imaging — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2001&filename=YXWZ200101009&uniplatform=NZKPT&v=lVYC_AMvNqB4o4X1tQ7L22y6HQGl7QDAAN-b_0AR5SZ-brjNXnUXclpt3iEgQyuQ
- See also: Noninvasive monitoring of hypertensive intracerebral hemorrhage and perihematomal tissue edema — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2003&filename=ZHYX200306008&uniplatform=NZKPT&v=CAr8b2wwr3b7L8O8NxFHAC2KFXMdVrX51LitXvBPRsgejq8CVaMuVgwKAK8QInbv
- See also: Application of noninvasive cerebral electrical impedance measurement on brain edema in patients with intracerebral hemorrhage — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2007&filename=ZHSJ200706007&uniplatform=NZKPT&v=rxlfgEeP_kUAcTBIbfqYfRPuuVNEEzR8G9G4CfqzrNblOUph8Lyhw1BDdd6rlNpd
- See also: A new method of noninvasive brain-edema monitoring in patients with intracranial tumor: cerebral electrical impedance measurement — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CMFD&dbname=CMFD2010&filename=2010015764.nh&uniplatform=NZKPT&v=DZRsncyRWA-kDLE22rWY3SxXwHUbJSHInOPpMy4EgV2S9hjIL3368SpaJS0wzZ_N
- See also: An applied research on non-invasive and dynamic monitor of cerebral edema in patients after craniotomy — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2011&filename=LXYB201103016&uniplatform=NZKPT&v=pBUGsByuDjfeeKsmumQdEjnXla7Ybu3xGwem1DHVPYsNvIFvVN6_9ZbGPG2T4Gyd
- See also: Application of continuous intracranial pressure monitoring in hypertensive cerebral hemorrhge — https://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFD2012&filename=ZWQX201208005&uniplatform=NZKPT&v=qSCtlduJ1C_UjPQ_SJCYNecS2t62VxY_NmKKhHtDKo_LVmcFT8FYVnJJ2JKxP-cz